CLINICAL TRIAL: NCT04150536
Title: An Open Label, Randomized, Three-treatment, Three-sequence, Three-period, Cross-over, Pharmacokinetic and Adhesion Performance Study of Lidocaine Patch 36 mg/Patch (1.8%) in Fasting, Healthy, Adult, Human Subjects, With Physical Exercise, Heat and Normal Conditions.
Brief Title: Pharmacokinetics and Adhesion of Lidocaine Topical System 1.8% Under Conditions of Heat and Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SCI-LIDO-HEX-001
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lidocaine Topical System with Moderate Exercise (Treatment A) (Experimental): Three lidocaine topical systems 1.8% are applied to mid-lower back for 12 hours. Subjects are instructed to exercise 30 minutes on an exercise bicycle, achieving at heart rate of approximately 108 bpm. Exercise is performed after 2.5 hours, 5.5 hours, and 8.5 hours after topical system application.
  Interventions: Drug: Lidocaine topical system 1.8%
- Lidocaine Topical System with Heat Applied (Treatment B) (Experimental): Three lidocaine topical systems 1.8% are applied to mid-lower back for 12 hours. A heating pad is applied for 20 minutes at 2.5, 5.5, and 8.5 hours after the product is applied.
  Interventions: Drug: Lidocaine topical system 1.8%
- Lidocaine Topical System under normal conditions (Treatment C) (Experimental): Three lidocaine topical systems 1.8% are applied to mid-lower back for 12 hours. No heat application or exercise is performed during this period.
  Interventions: Drug: Lidocaine topical system 1.8%

INTERVENTIONS:
Drug: Lidocaine topical system 1.8%
  Other Names: ZTlido; Lidocaine patch 1.8%

SUMMARY:
The objectives of this study are to evaluate the pharmacokinetic and adhesion performance of ZTlido (lidocaine topical system) 1.8% during physical exercise, application of heat, and under normal conditions.

DETAILED DESCRIPTION:
In this open-label, three-period crossover study, 12 healthy, adult male and female subjects are randomized to 1 of 3 treatment sequences. During each treatment period, subjects have three lidocaine topical systems applied to their back for 12 hours with 7-day washout between treatments. In each treatment period, the subject will either exercise (Treatment A), apply a heating pad (Treatment B), or refrain from these activities (Treatment C) while wearing the topical system. Blood samples for lidocaine PK will be collected pre-dose until 48 hours. Adhesion will be monitored throughout the wear time and skin irritation will be assessed the topical system is removed.

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on by medical history, laboratory work, and physical exam
* Be at least 18 years of age
* If childbearing potential, use of acceptable form of birth control
* In the case of females of childbearing potential, have a negative serum pregnancy test

Key Exclusion Criteria:

* Allergy or known hypersensitivity to lidocaine, amide-type local anesthetics, or any component of the product formulation
* Any major medical illness 3 months prior or any significant history or ongoing chronic medical illness affecting the major body systems, including the skin
* Subjects with conditions that might affect application of the product or its adhesive properties (including psoriasis, eczema, atopic dermatitis, damaged or irritated epidermal layer, and excessive hair or oil on the skin)
* History of addiction, abuse, and misuse of any drug
* Use of nicotine-containing products within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of lidocaine | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22 24 and 48 hours post-dose
  Peak plasma concentration of lidocaine after application of 3 patches for 12 hours
Area under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time 48 hours | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22 24 and 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to 48 hours of lidocaine in plasma
Area under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time Infinity | 0, 2, 4, 6, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22 24 and 48 hours post-dose
  Area under the plasma concentration versus time curve from 0 to infinite time of lidocaine in plasma
Cumulative Adhesion Score | 0, 0.5, 3, 6, 9, 12 hours post-dose
  Adhesion to skin assessed by FDA 0-4 scoring system. The scoring for adhesion of patches is indicated as follows: 0 = ≥ 90% Adhered (essentially no lift off the skin), 1 = ≥ 75% to < 90% Adhered (some edges only lifting off the skin), 2 = ≥ 50% to < 75% Adhered (less than half of the patch lifting off the skin), > 0% to < 50% Adhered but not detached (more than half of the patch lifting off the skin without falling off), and 4 = 0% adhered (patched completely detached). The cumulative adhesion score is calculated as the sum of scores at each assessment time point.

SECONDARY OUTCOMES:
Dermal Response Score | 12.5 and 14 hours post-dose
  Product tolerability is assessed by Dermal Response Score. The application site is evaluated 30 minutes and 2 hours after product removal (12.5 and 14 hours post-dose, respectively). Response score from 0 to 7; 0= No evidence of irritation, 1= Minimal erythema, barely perceptible, 2= Definite erythema, readily visible; minimal edema or minimal papular response, 3= Erythema and papules, 4= Definite edema, 5= Erythema, edema and papules, 6= Vesicular eruption, 7= Strong reaction spreading beyond test (i.e., application) site.

CONTACTS AND LOCATIONS:
Overall Officials: John Peterson, PharmD, RPh, Principal Investigator — Axis Clinicals

REFERENCES:
- [Derived] Fudin J, Wegrzyn EL, Greuber E, Vought K, Patel K, Nalamachu S. A Randomized, Crossover, Pharmacokinetic and Adhesion Performance Study of a Lidocaine Topical System 1.8% During Physical Activity and Heat Treatment in Healthy Subjects. J Pain Res. 2020 Jun 10;13:1359-1367. doi: 10.2147/JPR.S238268. eCollection 2020. PMID 32606902